CLINICAL TRIAL: NCT05271253
Title: Comparison Between Different Anaesthesia Techniques for Protecting Renal Function in Children Undergoing Radicle Nephrectomy
Brief Title: Comparison Between Different Anaesthesia Techniques Protecting Renal Function in Children Undergoing Radicle Nephrectomy
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Alexandria University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 0305085
Record Dates: First submitted 2022-01-27; First posted 2022-03-09 (Actual); Last update posted 2022-03-09 (Actual); Status verified 2022-01

CONDITIONS: Renal Injury; Child, Only
Keywords: radical nephrectomy
MeSH Terms: interventions — Dexmedetomidine; Bupivacaine; Saline Solution; Sodium Chloride

STUDY DESIGN:
Intervention Model Description: Patients were randomly allocated into 3 equal groups (25 patients each): Group (C): caudal group, where caudal anaesthesia was given using 1 mL/kg dose of 0.25% bupivacaine without epinephrine. Dexmedetomidine (D) group, where Dex. (Precedex, hospira, Egypt) 0.8 μg/kg was given intravenously over 10 min as a loading dose, and then infused at a rate of 0.4 μg/kg/h; and Placebo (P) group, where normal saline instead of Dex was given in volume (ml) and rate (ml/h) calculated related to the patient's body weight.
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Group (C) (Active Comparator): caudal group, where caudal anaesthesia was given using 1 mL/kg dose of 0.25% bupivacaine without epinephrine.
  Interventions: Drug: bupivacaine
- Group (D) (Active Comparator): Dexmedetomidine (D) group, where Dex. (Precedex, hospira, Egypt) 0.8 μg/kg was given intravenously over 10 min as a loading dose, and then infused at a rate of 0.4 μg/kg/h
  Interventions: Drug: Dexmedetomidine
- Group (P) (Placebo Comparator): Placebo (P) group, where normal saline instead of Dex was given in volume (ml) and rate (ml/h) calculated related to the patient's body weight.
  Interventions: Drug: normal Saline

INTERVENTIONS:
Drug: Dexmedetomidine — 0.5 mic /kg dexmedetomedine is injected after induction of anaesthesia.
  Other Names: preceedex
  Arms: Group (D)
Drug: bupivacaine — 0.25% bupivacaine is injected in the caudal epidural space
  Arms: Group (C)
Drug: normal Saline — injection of normal Saline
  Other Names: 0.9 % Nacl
  Arms: Group (P)

SUMMARY:
Up to date, Renal Cell carcinomas (RCC) are one of the prevalent primary renal neoplasms affecting children & surgical radical nephrectomy is the conventional standard of care, as the choice of non-surgical modalities like irradiation & hormono-chemotherapy is still a subject of debate .

Worsening of postoperative renal function is not so far from these patients who underwent nephrectomy for RCC, thus peri-operative preservation of renal function is a great challenge facing anaesthologist aiming to abolishment of postoperative acute kidney injury (AKI) development. AKI is a serious clinical diverse which increases morbidity and mortality & enhances the risk of development of chronic kidney disease (CKD). A major advances have shown that the associations between AKI and CKD after radical nephrectomy is as high as 65 %.

For years, the diagnosis of AKI was based on ordinary kidney function tests like serum creatinine & blood urea nitrogen, which are not efficient nowadays, as they lack specificity for renal damage, besides they are affected by many other factors apart from kidney injury.

Cystatin C is an endogenous protein with low molecular weight (13 k Da), that is freely filtrated at the glomeruli and completely reabsorbed in the proximal renal tubules. It indicates renal injury indirectly through decreased GFR .

Serum neutrophil gelatinase-associated lipocalin (NGAL) is a promising glycoprotein produced by neutrophils and epithelial cells of the proximal convoluted tubule of the nephron cells. After renal stress or nephrotoxic damage its peak plasma level is reached within 6 hrs, then remains sustained for as long as 5 days.

Dexmedetomidine (Dex.) a newer, short acting, highly selective alph-2 agonist, that possess potent analgesic, amnestic, hypnotic & sedative properties via actions on sleep-awake cycle in the brain. Several evidences reported its possible ability for renal protection.

Caudal epidural blockade is well known efficient technique that offer postoperative analgesia for multiple surgical procedures in children. Beside hemodynamic stability, they prevent progression of acute postoperative pain to chronic pain.

The investigators hypothesized that uses of Dex infusion in a programmed fashion in children undergoing RN, could produce optimum preservation of kidney function from the concurrent perioperative insult even in a very early phase of renal stress, relative to ordinary used protocols.

DETAILED DESCRIPTION:
Aim of the study The primary goal was comparison between different anaesthesia techniques in preservation of kidney function using early phase detectors cystatin C and NGAL. Secondary goals included measurements of creatinine clearance, serum creatinine, and urinary output. Postoperative pain assessment using visual analogue scale & sedation score were also recorded.

3. Patients and methods

After approval of the Ethical committee of faculty of Medicine, Alexandria University and obtaining an informed written consent from parents of the children included in the study, 75 patients aged 5-10 years undergoing elective RN were randomly enrolled using closed envelope method. Sample Size was calculated according to the following equation:

n=(t^2×p(1-p))/m^3

The patients were excluded if they had history of use of α 2-agonists to treat hypertension, renal impairment (creatinine clearance < 90 ml/min), and persistent intraoperative hypotension [mean arterial blood pressure < 65 for > 20 min]. Also those with bleeding disorders and skin lesion at puncture site.

Patients were randomly allocated into 3 equal groups (25 patients each): Group (C): caudal group, where caudal anaesthesia was given using 1 mL/kg dose of 0.25% bupivacaine without epinephrine. Dexmedetomidine (D) group, where Dex. (Precedex, hospira, Egypt) 0.8 μg/kg was given intravenously over 10 min as a loading dose, and then infused at a rate of 0.4 μg/kg/h; and Placebo (P) group, where normal saline instead of Dex was given in volume (ml) and rate (ml/h) calculated related to the patient's body weight. The infusions were prepared by independent participant & were started after induction of anaesthesia and continued 24 hrs postoperatively. All children were assessed thoroughly preoperatively by history taking, physical examination & laboratory investigations (complete blood count, coagulation profile liver function & kidney functions.) At the night before surgery, base line value of serum creatinine, creatinine clearance were obtained using standard laboratory methods. Also, base line value of serum cystatin C and NGAL were obtained using commercially available kits (Roche Diagnostics, Mannheim, Germany) & (Biosite Incorporated, San Diego, CA, USA) respectively by ELISA method. Establishment of method and degree of sample dilution were carried out prior to analysis according to manufacture instruction.

All children were premedicated orally with midazolam 0.5 mg/ k.g 30 minutes before induction, and they were instructed to void just before admission to the operating room.

In the operating theater, all patients were monitored throughout surgery by continuous electrocardiography, heart rate, pulse oximetry, non invasive blood pressure and end tidal capnography by (Datex-Omeda model S/5) monitor. Induction was carried out with fentanyl (1-1.5 μg/kg), and propofol (1-2 mg/kg). For facilitating endotracheal intubation, atracurium was administered at an initial dose of 0.5 mg/kg followed by boluses of 0.03 mg/kg every 20-40 min. Under aseptic technique, an arterial line and central venous catheter were inserted & Anaesthesia was maintained using isoflurane 1-2% in oxygen, and patients were mechanically ventilated. Fentanyl and atracurium increments were given as required.

The diagnostic criteria of AKI was classified according to the Acute Kidney Injury Network (AKIN) criteria as follows: the renal function decreased rapidly within 48 hours, the s Cr level increased by ≥ 26.5 µ mol/L or ≥ 1.5 times from baseline, or urine output < 0.5 mL/kg/h for > 6 hours. Oliguria is defined as urine output < 0.5 ml/kg/h. After exclusion of catheter obstruction, patients were managed with good hydration. If it persists, 10 mg I.v Lasix was given, that could be repeated twice. If no response, nephrology consultation was ordered. At the end of surgery, muscle relaxants were reversed by neostigmine 0.04-0.06 mg/kg and atropine 0.02 mg/kg, and then the patients were extubated after returning to full muscle power. All patients were monitored in the intensive care unit for 2 days after surgery, with attention to fluid balance and urine output. Serum creatinine, creatinine clearance, Cystatin C and NGAL was assessed 24 hr before surgery, after induction of anaesthesia, 12 and 24 hrs postoperatively. Urine output was assessed intraoperatively every 1 hr and postoperatively every 6 hr in the first 24 hrs. Sedation was assessed during the first 5, 15, 30, and 60 mins in the recovery room by the investigator using a five-point sedation scale. Sedation level: Agitated = 4, Awake= 3, Drowsy= 2, Asleep= 1. A sedation score of 3 & above was considered as unsatistisfactory while 1&2 is considered to be satisfactory. Postoperative pain was assessed using the visual analog scale from 0-10, where 0= no pain and 10= unbearable pain.

Data management Data were fed to the computer and analyzed using IBM SPSS software package version 20.0 (Armonk, NY: IBM Corp). Quantitative data were described using range (minimum and maximum), mean, SD, and median. Significance of the obtained results was judged at the 5% level.

ELIGIBILITY:
Inclusion Criteria:

* patients aged 5-10 years undergoing elective RN

Exclusion Criteria:

* had history of use of α 2-agonists to treat hypertension, renal impairment (creatinine clearance < 90 ml/min), and persistent intraoperative hypotension [mean arterial blood pressure < 65 for > 20 min]. Also those with bleeding disorders and skin lesion at puncture site.

Ages: 5 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 75 (Actual)
Dates: Start 2021-04-10 (Actual); Primary Completion 2021-11-29 (Actual); Study Completion 2022-01-15 (Actual)

PRIMARY OUTCOMES:
cystatin C | immediately after induction
  Early biomarkers in detection of renal impairment
cystatin C | after 12 hours post-operatively
  Early biomarkers in detection of renal impairment
NGAL | immediately after induction
  Early biomarkers in detection of renal impairment
NGAL | after 12 hours post-operatively
  Early biomarkers in detection of renal impairment

SECONDARY OUTCOMES:
serum creatinine | immediately after induction
  conventional renal function tests
serum creatinine | after 12 hours post-operatively
  conventional renal function tests
creatinine clearance | immediately after induction
  conventional renal function tests
creatinine clearance | after 12 hours post-operatively
  conventional renal function tests
sedation score | 5 mins post-operative
  indicator for post operative alertness, . Sedation level: Agitated = 4, Awake= 3, Drowsy= 2, Asleep= 1. A sedation score of 3 & above was considered as unsatisfactory while 1 & 2 is considered to be satisfactory.
sedation score | 60 mins post-operative
  indicator for post operative alertness,. Sedation level: Agitated = 4, Awake= 3, Drowsy= 2, Asleep= 1. A sedation score of 3 & above was considered as unsatisfactory while 1 & 2 is considered to be satisfactory.

CONTACTS AND LOCATIONS:
Overall Officials: Hassan S ElHoshy, lecturer, Study Chair — Alexandria University
Locations (1):
- Haasan Elhoshy, Alexandria, Egypt

IPD SHARING:
Plan to Share IPD: No